CLINICAL TRIAL: NCT02385461
Title: A Proposal of a Prospective Study on Prevention of Pregnancy Loss in Women Carrying Inherited Thrombophilia
Brief Title: Study on Antithrombotic Prevention in Thrombophilia and Pregnancy Loss
Acronym: OTTILIA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Casa Sollievo della Sofferenza IRCCS (Other)
Responsible Party: Principal Investigator, Elvira Grandone, MD, Head of Unit, A proposal of a prospective study on prevention of pregnancy loss in women carrying inherited thrombophilia., Casa Sollievo della Sofferenza IRCCS
Other Study IDs: EMOST 01/2011
Record Dates: First submitted 2015-03-05; First posted 2015-03-11 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Pregnancy Complications
MeSH Terms: conditions — Pregnancy Complications | interventions — Dalteparin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Inherited Thrombophilia: Women with Common Inherited Thrombophilias and previous foetal loss
  Interventions: Drug: Low Molecular Weight Heparins (LMWHs)
- Other Thrombophilias with Pregnancy loss: Women with Thrombophilias other than common inherited thrombophilias and previous foetal loss
  Interventions: Drug: Low Molecular Weight Heparins (LMWHs)
- No thrombophilia: Women without thrombophilias and previous foetal loss
  Interventions: Drug: Low Molecular Weight Heparins (LMWHs)

INTERVENTIONS:
Drug: Low Molecular Weight Heparins (LMWHs)

SUMMARY:
The occurrence of a spontaneous fetal loss (FL) is a rather frequent event: it has been estimated that up to 15% of pregnancies result in a fetal loss. However, recurrent events, defined as >2 or >3 loss, depending on the guidelines used (American College of Obstetricians and Gynecologists or Royal College of Obstetricians Gynaecologists guidelines), occur in 1 % of all pregnancies and it is noteworthy that Recurrent Fetal Loss ( RFL) in about 30-40% of cases remain unexplained after standard gynaecological, hormonal and karyotype investigations. Furthermore, it is important to consider that chromosomal abnormalities are responsible for at least 60% of FL in the first trimester, thus an abnormal karyotype in the fetus should be excluded prior to consider testing women for genetic susceptibility to placental vascular complications (inherited thrombophilia).

Common inherited conditions, the factor V Leiden (FV) and the factor II G20210A (FII) mutations have been recognized as risk factors for FL.

The efficacy of treatment with antithrombotic drugs during pregnancy in women with a history of RFL/ Intra Uterine Fetal Death (IUFD) and thrombophilia is still debated, due to scarcity of available data. Italian guidelines suggest the use of Low-Molecular-Weight Heparin (LMWH) in women with FV or FII mutations and previous otherwise unexplained obstetric complications, while guidelines released by RCOG suggest that heparin therapy during pregnancy may improve the live birth rate in women with second trimester loss associated with inherited thrombophilias. Hence, the idea to propose this prospective observational study comparing clinical data and outcomes in women with common inherited thrombophilias and in women without.

During this study the investigators will collect and evaluate clinical data from examinations and visits by patients, eligible for the study as carriers of thrombophilic defects. This observation will begin before pregnancy and continue until the puerperium, allowing us to study all possible factors influencing these conditions. The study will add knowledge for improving feto-maternal prognosis and preventing spontaneous and recurrent FL.

Plan of the study: multicenter observational study

ELIGIBILITY:
Inclusion Criteria:

* recurrent otherwise unexplained FL (defined as >3, or 2 in the presence of at least 1 normal fetal karyotype) (according to Lussana et al.) or
* at least 1 intrauterine fetal death (IUFD), defined as a loss after 20 weeks of a morphologically normal fetus with/without HETEROZYGOUS FOR FACTOR V LEIDEN or HETEROZYGOUS FOR FIIA20210 (PTm)

Exclusion Criteria:

* personal history of venous and/or arterial thromboembolism;
* documented hemorrhagic disease;
* allergy to LMWH;
* uterine abnormalities;
* cervical incompetence;
* untreated endocrine diseases (diabetes mellitus or thyroid disease);
* indication to anticoagulant treatment during pregnancy;
* chromosomal abnormalities in parents

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Consecutive pregnant women with previous pregnancy loss
Sampling Method: Probability Sample
Enrollment: 108 (Estimated)
Dates: Start 2012-01; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Number of live births | 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Elvira Grandone, MD, Principal Investigator — Thrombosis Unit, I.R.C.C.S. Casa Sollievo della Sofferenza, S. Giovanni Rotondo (Foggia)
Locations (1):
- I.R.C.C.S. Casa Sollievo della Sofferenza, San Giovanni Rotondo, Foggia, Italy

REFERENCES:
- [Derived] Grandone E, Tiscia GL, Mastroianno M, Larciprete G, Kovac M, Tamborini Permunian E, Lojacono A, Barcellona D, Bitsadze V, Khizroeva J, Makatsarya A, Cacciola R, Martinelli I, Bucherini E, De Stefano V, Lodigiani C, Colaizzo D, De Laurenzo A, Piazza G, Margaglione M. Findings from a multicentre, observational study on reproductive outcomes in women with unexplained recurrent pregnancy loss: the OTTILIA registry. Hum Reprod. 2021 Jul 19;36(8):2083-2090. doi: 10.1093/humrep/deab153. PMID 34195794
- [Derived] Villani M, Baldini D, Totaro P, Larciprete G, Kovac M, Carone D, Passamonti SM, Permunian ET, Bartolotti T, Lojacono A, Cacciola R, Pinto GL, Bucherini E, De Stefano V, Lodigiani C, Lavopa C, Cho YS, Pizzicaroli C, Colaizzo D, Grandone E. Rationale and design of two prospective, multicenter, observational studies on reproductive outcome in women with recurrent failures after spontaneous or assisted conception: OTTILIA and FIRST registries. BMC Pregnancy Childbirth. 2019 Aug 13;19(1):292. doi: 10.1186/s12884-019-2444-y. PMID 31409287